CLINICAL TRIAL: NCT04054908
Title: Gut Microbiome and Oral Fluoropyrimidine Study in Patients With Colorectal Cancer
Brief Title: Gut Microbiome in Colorectal Cancer
Acronym: GO
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 174527; R21CA227232 (NIH)
Record Dates: First submitted 2019-07-18; First posted 2019-08-13 (Actual); Last update posted 2024-06-14 (Actual); Status verified 2022-09

CONDITIONS: Gastrointestinal Microbiome; Neoplasm, Colorectal
Keywords: Gut Microbiome; Colorectal Cancer; Oral Fluoropyrimidine
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Stool samples will be collected from patient over course of the standard of care for colorectal cancer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Cohort A: Patients treated with oral fluoropyrimidine (Capecitabine (CAP)) as part of standard of care (SOC) chemotherapy
- Cohort B: Patients treated with Trifluridine/Tipiracil (TAS-102) including those receiving it in combination with Y-90 radioembolization as part of a clinical trial
- Cohort C: Patients receiving CAP plus immunotherapy (pembrolizumab) and bevacizumab as part of a clinical trial.

SUMMARY:
This is a pilot feasibility study designed to investigate the alterations in the gut microbiome that occur during the course of treatment for colorectal cancer

DETAILED DESCRIPTION:
This is a pilot feasibility study designed to investigate the alterations in the gut microbiome that occur during the course of treatment for colorectal cancer (CRC). Three patient cohorts will be followed. Cohort A: patients treated with oral fluoropyrimidine CAP as part of standard of care (SOC) chemotherapy. Cohort B: patients treated with TAS-102 including those receiving it in combination with Y-90 radioembolization as part of a clinical trial. Cohort C: patients receiving CAP plus immunotherapy (pembrolizumab) and bevacizumab as part of a clinical trial. Investigators will replace participants as needed to ensure a minimum of 10 evaluable participants per cohort (or minimum total of 30 evaluable patients). Evaluable participants are defined as patients with two analyzable stool samples including a baseline sample and at least one on-treatment sample to be used in endpoint analysis

ELIGIBILITY:
Inclusion Criteria:

1. The patient has histologically proven colorectal adenocarcinoma
2. The patient is starting treatment with oral fluoropyrimidine therapy: CAP or TAS-102 as SOC or on a clinical trial. This also includes those patients receiving treatment in the adjuvant setting or post-metastasectomy with no evidence of disease on imaging.
3. Combination of oral fluoropyrimidine with other cancer-directed therapies, including oxaliplatin, bevacizumab, Y-90 radioembolization, or immunotherapy checkpoint inhibitors, is permitted.
4. Combination of CAP with concurrent radiation is permitted, including patients undergoing radiotherapy to a rectal primary or a metastatic site.
5. Male or female patient aged 18 years of age or older at the time of obtaining the signed and dated informed consent (no upper age limit).
6. Be able to read and speak English.
7. Be willing and able to provide written informed consent for the study

Exclusion Criteria:

1. Patient has had prior chemotherapy, biologic or immunotherapy in the previous 2 weeks.
2. Patient has completed a course of antibiotics longer than 2 weeks in preceding six months or a course of antibiotics of any duration in the 4 weeks prior to starting oral chemotherapy. Any patient who requires treatment with antibiotics during the study may be removed at the investigator's discretion.
3. Known HIV positive.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recruitment will include both patients who will be taking TAS-102 and those taking CAP with or without other cancer-directed therapies, including those receiving CAP in combination with concurrent rectal radiation. Patients with colorectal cancer (CRC) expected to receive CAP or TAS-102 will be screened by the study PI, co-investigators, or study coordinators. The study coordinator may identify potential participants by various mechanisms: direct referral from a treating physician, review of schedules of medical and oncology providers at UCSF and participating sites, or phone calls from patients or referring physicians.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-04-13 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Recruitment rate rate (percentage of patients approached that consent to participate) | Up to 2 years
  Feasibility and acceptability will be assessed by evaluating percentage of patients approached that consent to participate
Reasons for nonparticipation/non-continuation of the study and adherence of submission of stool specimens | Up to 2 years
  Feasibility and acceptability will be assessed by evaluating reasons for nonparticipation/non-continuation of the study and adherence of submission of stool specimens
Dietary Assessment Questionnaires | Baseline, Day 1, Day 3, Day 7, Day 14, Day 21, at discontinuation of treatment (an average of 6 months)
  Baseline questionnaires regarding bowel habits and dietary history. Patients will complete a 3-day diet record (Automated SelfAdministered 24-Hour (ASA24®) Dietary Assessment Tool or on paper) at the beginning of each treatment cycle when stool is collected. For mid-cycle or toxicity-related stool collections, patients will complete a 24-hour diet recall using the ASA24 system
Acceptability of specimens for analysis | Up to 6 months
  Specimens collected via Fecal occult blood test (FOBT) card method will be verified as evaluable defined as patients with two analyzable stool samples including a baseline sample and at least one on-treatment sample to be used in endpoint analysis.

SECONDARY OUTCOMES:
Change in gut microbiome diversity | Up to 2 years
  Changes in the gut microbiome will be assessed by comparing the bacterial diversity present in the baseline pre-treatment stool sample to the designated initial treatment cycle midpoint for each of the three patient cohorts
Change in relative abundance of following gut bacteria that occur with oral fluoropyrimidine therapy | Up to 2 years
  Changes in relative and absolute abundance of specific bacteria from the Fusobacterium and Porphyromonas genus, and the species Bacteroides fragilis will be assessed using quantitative polymerase chain reaction (qPCR) and genus-specific primers

CONTACTS AND LOCATIONS:
Overall Officials: Wesley Kidder, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be shared with researchers at other institutions.

DOCUMENTS (1):
  • Informed Consent Form (2021-11-16): https://cdn.clinicaltrials.gov/large-docs/08/NCT04054908/ICF_000.pdf